CLINICAL TRIAL: NCT03644511
Title: Use of Sorafenib and/or Regorafenib in Hepatocellular Carcinoma (HCC) Subsequent to Another Systemic First-line Treatment
Brief Title: Use of Sorafenib and/or Regorafenib in Liver Cancer (Hepatocellular Carcinoma) Subsequent to Another Systemic First-line Treatment
Acronym: SORAGO-HCC
Status: Terminated | Type: Observational
Why Stopped: The interest of potential centers is very limited.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20215
Record Dates: First submitted 2018-08-22; First posted 2018-08-23 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; Liver cancer; Live cell carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — regorafenib; Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HCC: Treated with Nexavar and/or Stivarga as ≥ 2nd-line systemic treatment
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506); Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Prescribed by physician.
Drug: Sorafenib (Nexavar, BAY43-9006) — Prescribed by physician.

SUMMARY:
Researchers already did trials that showed Sorafenib and Regorafenib worked for patients with hepatocellular carcinoma (most common liver tumor type).

In this trial, they want to learn more about the same patient group in which Sorafenib or Regorafenib is given after other drugs. Patients participating in this study will be observed until 12 months after the last patient has been enrolled to collect data on how safe the drugs are and how well they are working when used as second line or beyond treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatocellular cancer in stage BCLC-B or BCLC-C
* Decision to initiate treatment with Nexavar (sorafenib) and/or Stivarga (regorafenib) as 2nd-line or beyond treatment was made as per investigator's routine treatment practice. Stivarga (regorafenib) must be used according to its indication, i.e. after prior progression under Nexavar (sorafenib) treatment.

Exclusion Criteria:

* Patients concurrently participating in an investigational program for the treatment of HCC with interventions outside of routine clinical practice.
* Stivarga (regorafenib) treatment without prior therapy with Nexavar (sorafenib). NOTE: Nexavar (sorafenib) treatment could have been given as treatment for HCC outside of this non-interventional study. In this case Stivarga (regorafenib) would NOT constitute the second-line therapy after direct pretreatment with Nexavar (sorafenib) but e.g. 3rd-line treatment directly after a different drug.
* Contra-indications according to the local marketing authorization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with HCC in stage BCLC-B (Barcelona Classification of Liver Cancer) or BCLC-C for whom the decision to treat with Nexavar and/or Stivarga as ≥ 2nd-line has been taken by the investigator and the drugs are prescribed in the customary manner in accordance with the terms of the marketing authorization.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Identification of current treatment patterns by means of individual treatment lines in the systemic HCC therapy with regards to Nexavar and Stivarga, i.e. when both drugs are used in ≥ 2nd-line under current practice conditions | Up to 24 months

SECONDARY OUTCOMES:
Overall Survival (OS) from start of Nexavar or Stivarga therapy and from start of first systemic therapy | Up to 36 months
Progression free survival (PFS) | Up to 36 months
Time to progression (TTP) | Up to 36 months
Duration of Nexavar or Stivarga treatment | Up to 36 months
Tumor response to treatment | Up to 36 months
  Evaluated by the investigator according to the categories "complete response", "partial response", "stable disease", "progressive disease by clinical judgment", "progressive disease measurement proven", "unknown" and "not applicable", and will be analyzed providing absolute and relative frequencies of the tumor status categories.
Incidence of treatment-emergent adverse events (TEAE) | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.